CLINICAL TRIAL: NCT05688904
Title: Pilot Studies Testing the Effect of Topical Imipramine on Pain and Effectiveness of Topical Photodynamic Therapy
Brief Title: The Effect of Topical Imipramine on Pain and Effectiveness of Topical Photodynamic Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 07286
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Imipramine; Photodynamic Therapy; Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Imipramine (Active Comparator): Topical 4% Imipramine
  Interventions: Drug: Imipramine
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Imipramine — Topical 4% Imipramine
  Arms: Imipramine
Other: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is testing the use of topical Imipramine in combination with topical photodynamic therapy's (PDT) effect on pain following treatment. PDT is a commonly used treatment in dermatology for patients who have many pre-cancers (actinic keratosis-AKs) on their skin. These are both FDA-approved treatments, but this study is evaluating their use in combination, which has not been evaluated in the past. The investigators have been doing studies using animals that suggest that imipramine might make the PDT less painful and might help it work better. In order to participate, the subject and their dermatologist have decided that they would benefit from PDT to treat their skin due to many AK precancerous lesions. Please note that neither PDT nor imipramine are experimental treatments, but treating their skin with imipramine before PDT is a new approach.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 and older
* Skin type must be "Fair", Fitzpatrick type I to III, due to the presence of actinic damage in this population.
* Subjects need to have a physician's order to receive PDT treatment on their face, scalp or forearms.
* Willing to participate and understand the informed consent document.
* Willing to avoid excess sun exposure/tanning beds to the area to be treated with PDT.

Exclusion Criteria:

* Those currently taking any tricyclic antidepressants (TCAs)
* Those currently taking any selective serotonin reuptake inhibitor (SSRI)
* Those with porphyria
* Large tattoos in the treated areas
* Pregnancy or nursing
* Taking any oral or topical medications that could interfere with the PDT (Appendix A)
* Active rashes in the area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of precancerous actinic keratosis present from baseline. | 6 months post PDT treatment
  Principal investigator assesses this from AK lesion count mapping at baseline and in 6 months.

SECONDARY OUTCOMES:
Change in pain level due to photodynamic therapy (PDT) from baseline. | Immediately post PDT treatment
  The visual analog pain scale is used to assess this outcome. (0 = no skin pain to 10 = severe skin pain)
Change in pain level due to photodynamic therapy (PDT) from baseline. | 10 minutes post PDT treatment
  The visual analog pain scale is used to assess this outcome. (0 = no skin pain to 10 = severe skin pain)
Change in pain level due to photodynamic therapy (PDT) from baseline. | 30 minutes post PDT treatment
  The visual analog pain scale is used to assess this outcome. (0 = no skin pain to 10 = severe skin pain)
Change in pain level due to photodynamic therapy (PDT) from baseline. | 6 months post PDT treatment
  The visual analog pain scale is used to assess this outcome. (0 = no skin pain to 10 = severe skin pain)
Change in itch level due to photodynamic therapy (PDT) from baseline. | Immediately post PDT treatment
  The visual analog itch scale will be used to assess this outcome. (0 = no skin itch to 10 = severe skin itch)
Change in itch level due to photodynamic therapy (PDT) from baseline. | 10 minutes post PDT treatment
  The visual analog itch scale will be used to assess this outcome. (0 = no skin itch to 10 = severe skin itch)
Change in itch level due to photodynamic therapy (PDT) from baseline. | 30 minutes post PDT treatment
  The visual analog itch scale will be used to assess this outcome. (0 = no skin itch to 10 = severe skin itch)
Change in itch level due to photodynamic therapy (PDT) from baseline. | 6 months post PDT treatment
  The visual analog itch scale will be used to assess this outcome. (0 = no skin itch to 10 = severe skin itch)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Rohan, MD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT05688904/ICF_000.pdf